CLINICAL TRIAL: NCT04040712
Title: Fecal Microbiota Transplantation to Treat Diarrhea Induced by Tyrosine-kinase Inhibitors in Patients With Metastatic Renal Cell Carcinoma: a Randomized Clinical Trial.
Brief Title: Fecal Microbiota Transplantation in Diarrhea Induced by Tyrosine-kinase Inhibitors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Giovanni Cammarota, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMT-TKI-001
Record Dates: First submitted 2019-04-22; First posted 2019-08-01 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Diarrhea Caused by Drug (Disorder); Renal Cell Cancer
Keywords: fecal microbiota transplantation; microbiota; chemotherapy; diarrhea; renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donor FMT (Experimental): Fecal microbiota transplantation using stools from healthy donors
  Interventions: Other: Donor FMT
- Sham FMT (Sham Comparator): Sham fecal microbiota transplantation
  Interventions: Other: Sham FMT

INTERVENTIONS:
Other: Donor FMT — Fecal microbiota transplantation using stools from healthy donors
  Arms: Donor FMT
Other: Sham FMT — Sham fecal microbiota transplantation
  Arms: Sham FMT

SUMMARY:
Tyrosine kinase inhibitors (TKIs) have improved the survival of patients with metastatic renal cell carcinoma, and are commonly used as first-line option for this condition, but their use is encumbered by side effects, mainly diarrhea, for which there are no standardized strategies. Increasing evidence suggests that gut microbiota could influence the development of TKIs-induced diarrhea. In theory, the therapeutic modulation of gut microbiota could be an approach to alleviate TKI-induced diarrhea. Fecal microbiota transplantation (FMT) is the infusion of fecal microbiota from a healthy donor in the gut of a recipient with the aim of curing a specific disease. It has been increasingly recognized as a highly effective treatment against recurrent Clostridium difficile infection.To date, the effects of FMT on chemotherapy-related diarrhea are unknown. This study will evaluate, through a randomized controlled design, the efficacy of fecal microbiota transplantation (FMT), compared with sham FMT, in treating TKI-induced diarrhea in patients with metastatic renal cell carcinoma.

DETAILED DESCRIPTION:
Despite the improvement in diagnosis and management, renal cell carcinoma (RCC) remains one of the most burdensome urological cancers, being the sixth most common malignancy in men and the 10th in women, accounting, respectively, for 5% and 3% of all cancers. Moreover, the incidence of RCC is increasing, especially in Western countries, accounting for nearly 60000 new cases per year in the United States. A considerable proportion of patients present with metastatic disease at diagnosis, and there are more than 140000 RCC-dependent deaths per year worldwide according to the World Health Organization.

Sunitinib and pazopanib are oral multi-targeted receptor tyrosine kinase inhibitors (TKIs) that have dramatically improved the survival of patients with metastatic RCC, and are commonly used as first-line option for this condition.

However, long-term use of these drugs is prevented by the development of toxicity. Diarrhea is one of the most common side effects of TKIs, occurring in nearly 50% of patients. It decreases the quality of life of these patients, and often requires dose reduction and drug discontinuation, potentially decreasing the efficacy of TKIs.

To date there are no standardized strategies for TKIs-related diarrhea, and current recommendations are supported by few evidence or real-life experience. Recommended treatment options include anti-motility agents, which are not targeted to act on the pathogenic pathways of diarrhea.

Increasing evidence suggests that gut microbiota could influence the development of TKIs-induced diarrhea. Overall, chemotherapy is known to drive, through the development of mucositis, deep compositional and functional alterations of gut microbiota. Mucositis occurs commonly after treatment with TKIs, and a specific dysbiotic profile has been found in patients with TKIs-induced diarrhea.

In theory, the therapeutic modulation of gut microbiota could be an approach to alleviate TKI-induced diarrhea. Although probiotics have been suggested as a possible treatment option for this condition, few evidence supports this indication.

Fecal microbiota transplantation (FMT) is the infusion of fecal microbiota from a healthy donor in the gut of a recipient with the aim of curing a specific disease. It has been increasingly recognized as a highly effective treatment against recurrent Clostridium difficile infection.

FMT has been also examined as a potential approach for other disorders associated with a disruption of gut microbiota, including ulcerative colitis or metabolic syndrome.

To date, the effects of FMT on chemotherapy-related diarrhea are unknown. The aim of this study is to investigate the efficacy of fecal microbiota transplantation (FMT), compared with sham FMT, in treating TKI-induced diarrhea in patients with metastatic RCC

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* treatment with pazopanib or sunitinib for metastatic RCC diagnosed at histology and measurable according to RECIST criteria version 1.1
* development of diarrhea of 2-3 grade according to Common Terminology Criteria (CTC) for Adverse Events (AE) version 4.0 induced by these drugs.
* execution of a CT scan no earlier than 4 weeks before enrollment
* good or intermediate prognostic assessment (according to criteria of the prognostic system of the International Metastatic RCC Database Consortium)
* performance status equal or lower than 2
* blood count, hepatic and kidney testing within normal limit
* ability to give their consent to be included in the study.

Exclusion criteria:

* another known cause of diarrhea (e.g. infectious gastroenteritis. Clostridium difficile infection, celiac disease, inflammatory bowel disease, irritable bowel syndrome, chronic pancreatitis, biliary salt diarrhea)
* previous colorectal surgery or cutaneous stoma
* food allergies
* recent (<6 weeks) therapy with drugs that could possibly alter gut microbiota (e.g. antibiotics, probiotics, proton pump inhibitors, immunosuppressants, metformin)
* another cancer (except for surgically treated basocellular carcinoma)
* brain metastases
* decompensated heart failure or heart disease with ejection fraction lower than 30%
* severe respiratory insufficiency
* psychiatric disorders
* pregnancy
* unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2020-01-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
rate of patients who experience resolution of diarrhea 4 weeks after the end of treatments | 4 weeks
  rate of patients who experience resolution of diarrhea 4 weeks after the end of treatments

SECONDARY OUTCOMES:
rate of patients who need to stop or reduce treatment with tyrosine-kinase inhibitors | 4 weeks
  rate of patients who need to stop or reduce treatment with tyrosine-kinase inhibitors
rate of patients who experience resolution of diarrhea 1 week after the end of treatments | 1 week
  rate of patients who experience resolution of diarrhea 1 week after the end of treatments
rate of patients who experience resolution of diarrhea 2 weeks after the end of treatments | 2 weeks
  rate of patients who experience resolution of diarrhea 2 weeks after the end of treatments
rate of patients who experience resolution of diarrhea 8 weeks after the end of treatments | 8 weeks
  rate of patients who experience resolution of diarrhea 8 weeks after the end of treatments
rate of patients who experience decrease of diarrhea until grade G1 or lower 1 week after the end of treatments | 1 week
  rate of patients who experience decrease of diarrhea until grade G1 or lower 1 week after the end of treatments
rate of patients who experience decrease of diarrhea until grade G1 or lower 2 weeks after the end of treatments | 2 weeks
  rate of patients who experience decrease of diarrhea until grade G1 or lower 2 weeks after the end of treatments
rate of patients who experience decrease of diarrhea until grade G1 or lower 4 weeks after the end of treatments | 4 weeks
  rate of patients who experience decrease of diarrhea until grade G1 or lower 4 weeks after the end of treatments
rate of patients who experience decrease of diarrhea until grade G1 or lower 8 weeks after the end of treatments | 8 weeks
  rate of patients who experience decrease of diarrhea until grade G1 or lower 8 weeks after the end of treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario "A. Gemelli" IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ianiro G, Rossi E, Thomas AM, Schinzari G, Masucci L, Quaranta G, Settanni CR, Lopetuso LR, Armanini F, Blanco-Miguez A, Asnicar F, Consolandi C, Iacovelli R, Sanguinetti M, Tortora G, Gasbarrini A, Segata N, Cammarota G. Faecal microbiota transplantation for the treatment of diarrhoea induced by tyrosine-kinase inhibitors in patients with metastatic renal cell carcinoma. Nat Commun. 2020 Aug 28;11(1):4333. doi: 10.1038/s41467-020-18127-y. PMID 32859933